CLINICAL TRIAL: NCT00661596
Title: Multi-centre, Randomised, Double-blind, Parallel, Placebo-controlled Clinical Study to Assess the Efficacy of Vardenafil and Its Influence on Self-esteem and Self-confidence in Patients With Erectile Dysfunction
Brief Title: Assessment of Efficacy of Vardenafil, Influence on Self-esteem and Self-confidence in Subjects With Erectile Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11139
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Vardenafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — 5 mg, 10 mg and 20 mg one hour prior to sexual intercourse
  Arms: Arm 1
Drug: Placebo — Matching placebo
  Arms: Arm 2

SUMMARY:
Erectile problems may lead to anxiety, loss of self-esteem and depression and/or stress. The purpose of this national study was to determine if vardenafil is effective in treating impotent men (erectile dysfunction) and evaluate its influence in self-esteem and self-confidence. During the visits the patients was asked some questions about erections, and he fill different questionnaires about sexuality, mood, feelings, self-esteem and sexual activity.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and older
* Males with erectile dysfunction
* Stable heterosexual relationship

Exclusion Criteria:

* Primary hypoactive sexual desire- History of myocardial infarction, stroke or life-threatening arrhythmia within the prior 6 months
* Nitrate use
* Other exclusion criteria apply acc. to Summary of Product Characteristics

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2003-05; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
International Index of Erectile Function - Erectile Function Domain | 12 weeks

SECONDARY OUTCOMES:
Global Assessment Questionnaire | 12 weeks
IIEF-EF domain score | 12 weeks
Other diary based variables | 12 weeks
Safety and tolerability | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (13):
- Spain (13):
  - Alicante, Alicante
  - Sabadell, Barcelona
  - Barcelona, Catalonia
  - Granada, Granada
  - Hondarribia, Guipuzcoa
  - Leganés, Madrid
  - Móstoles, Madrid
  - Málaga, Málaga
  - Vigo, Pontevedra
  - Oviedo, Principality of Asturias
  - Seville, Sevilla
  - Valencia, Valencia
  - Valladolid, Valladolid